CLINICAL TRIAL: NCT07089277
Title: External Validation of the Glasgow-Blatchford Bleeding Score in a Tunisian Population
Status: Recruiting | Type: Observational
Sponsor: Hôpital Universitaire Sahloul (Other)
Responsible Party: Principal Investigator, Riadh Boukef, Riadh Boukef, Hôpital Universitaire Sahloul
Other Study IDs: UGIB
Record Dates: First submitted 2025-04-24; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-05

CONDITIONS: Upper Gastrointestinal Bleeding (UGIB); Glasgow-Blatchford Score
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients consulting with Upper gastrointestinal bleeding: consulting ED with UGIB

SUMMARY:
This study aims to externally validate the Glasgow-Blatchford Score (GBS) in a Tunisian population presenting with non-traumatic upper gastrointestinal bleeding. Despite advances in endoscopic management, early risk stratification remains essential to guide clinical decision-making. In Tunisia, the routine hospitalization of all patients for observation presents a challenge, highlighting the need for reliable prognostic tools.

The study is designed as a multicenter, descriptive, and analytical investigation across several emergency departments. Adult patients (≥16 years) will be included, with follow-up conducted at 30 days to assess for adverse outcomes including rebleeding, the need for hemostasis, complications, and mortality.

Clinical and epidemiological data will be collected using a standardized form. Statistical analysis will evaluate the predictive performance of the GBS, focusing on sensitivity, specificity, and predictive values for 30-day outcomes.

The results are expected to determine whether GBS is a valid and useful tool for risk assessment in the Tunisian context, potentially aiding in more efficient and targeted patient management.

DETAILED DESCRIPTION:
Introduction:

Acute gastrointestinal bleeding is a common reason for emergency department visits and is associated with significant morbidity and mortality. The emergency physician plays a crucial role in rapid diagnosis, risk stratification, and appropriate management [1]. Although the incidence of gastro-duodenal ulcers has decreased in recent years, they remain the most frequent cause of upper gastrointestinal bleeding [2].

Diagnostic and therapeutic approaches have significantly improved, particularly with the wider availability of endoscopy. However, early assessment of bleeding severity and prognostic risk remains essential in patient management. Several prognostic scoring systems have been proposed, but few have been validated or widely adopted in clinical practice [2].

In Tunisia, as in many developing countries, a major challenge is the routine hospitalization of all patients for monitoring, although only a subset will develop complications. The use of prognostic scores such as the Glasgow-Blatchford Score could allow for better identification of at-risk patients and more targeted therapeutic strategies [3-4].

The Glasgow-Blatchford Score (GBS) is a widely used predictive tool for assessing the risk of severe complications in patients with upper gastrointestinal bleeding. However, its performance and validity have been minimally studied in the Tunisian population. This study aims to validate the Glasgow-Blatchford Score in a Tunisian cohort to confirm its relevance and utility in a local clinical context [5-7].

Objective:

The objective of this study is to perform an external validation of the Glasgow-Blatchford Score in a Tunisian population. We aim to assess its ability to predict adverse outcomes such as rebleeding, the need for hemostatic intervention, complications, and 30-day mortality.

Materials and Methods:

This will be a multicenter, descriptive, and analytical study conducted in the emergency departments of several hospitals in Tunisia. Patients included in the study will have presented to the emergency department with non-traumatic upper gastrointestinal bleeding.

Inclusion Criteria:

Adult patients (≥16 years) presenting with non-traumatic upper gastrointestinal bleeding.

Exclusion Criteria:

Patients under 16 years of age.

Diagnosis of external hemorrhoids with mucosal lesions.

Patients who do not consent, are lost to follow-up, or have incomplete data.

All patients must provide informed consent to participate in the study, and confidentiality will be maintained in accordance with ethical principles in clinical research.

Methodology:

Patient clinical data will be collected using a structured data collection form, which will include the Glasgow-Blatchford Score criteria along with epidemiological and clinical characteristics. Patients will be followed up via telephone on Day 30 to record any adverse events (rebleeding, need for hemostatic therapy, complications, and death).

Statistical Analysis:

Data will be entered and analyzed using SPSS version 26.0. The performance of the Glasgow-Blatchford Score will be assessed in terms of sensitivity, specificity, positive and negative predictive values, and its ability to predict 30-day mortality and complications.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) presenting with non-traumatic upper gastrointestinal bleeding

Exclusion Criteria:

* patients under 18 years of age.

Diagnosis of external hemorrhoids with mucosal lesions.

Patients who do not consent, are lost to follow-up, or have incomplete data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included in the study will have presented to the emergency department with non-traumatic upper gastrointestinal bleeding.
  Inclusion Criteria:
  Adult patients (≥16 years) presenting with non-traumatic upper gastrointestinal bleeding.
  Exclusion Criteria:
  Patients under 16 years of age.
  Diagnosis of external hemorrhoids with mucosal lesions.
  Patients who do not consent, are lost to follow-up, or have incomplete data.
  All patients must provide informed consent to participate in the study, and confidentiality will be maintained in accordance with ethical principles in clinical research.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
adverse outcomes such as rebleeding, the need for hemostatic intervention, complications and mortality at 30 days | 30 days
  adverse outcomes such as rebleeding, the need for hemostatic intervention, complications and mortality at 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Sahloul University Hospital, Sousse, Tunisia

IPD SHARING:
Plan to Share IPD: No